CLINICAL TRIAL: NCT01910116
Title: Treatment Efficacy of 'Shinbaro Capsule' in the Treatment of Hand Osteoarthritis: Randomized, Double-blinded, Placebo-controlled, Multicenter Investigator Initiated Trial.
Brief Title: Efficacy of Shinabro in Hand Osteoarthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Green Cross Corporation (Industry)
Responsible Party: Principal Investigator, Eun Bong Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GC6102F
Record Dates: First submitted 2013-07-22; First posted 2013-07-29 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-08

CONDITIONS: Hand Osteoarthritis
Keywords: osteoarthritis; hand; Shinbaro; GCSB-5
MeSH Terms: conditions — Osteoarthritis | interventions — shinbaro

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo 2 capsules, twice daily, for 12 weeks.
  Interventions: Drug: Placebo
- Shinbaro (Active Comparator): Shinbaro, 2 capsules (300mg), twice daily, for 12 weeks
  Interventions: Drug: Shinbaro

INTERVENTIONS:
Drug: Shinbaro — GCSB-5 (Shinbaro) is a mixture of six purified oriental herb extracts in a fixed ratio, namely, Saposhnikovia divaricata Schischk, Glycine max Merrill, Cibotium barometz J. Smith, Eucommia ulmoides Oliver, Achyranthes japonica Nakai, and Acanthopanax sessiliflorus Seem
  Other Names: GCSB-5
  Arms: Shinbaro
Drug: Placebo — The study medication and placebo were identical in appearance.
  Arms: Placebo

SUMMARY:
GCSB-5 ("Shinbaro capsule"), is a mixture of 6 oriental herbs that have anti-inflammatory and analgesic effects along with an excellent safety profile. This study is aimed at investigating efficacy of Shinbaro in the treatment of hand osteoarthritis which needs a long term treatment in a placebo controlled, double-blind randomized trial.

DETAILED DESCRIPTION:
Osteoarthritis (OA) as a common musculoskeletal disease affects more than 30% of the elderly population. It frequently involves knees, hips, spines and hands. In hands, the distal and proximal interphalangeal and the first carpometacarpal joints are affected, leading often to significant disability and limitation in the daily activity. The chronic progressive nature of the disease requires a life-long treatment. The mainstay treatment of hand OA targets pain control. Non-steroidal anti-inflammatory drugs (NSAIDs) are often used. However, they are frequently associated with significant gastrointestinal side effects including gastritis, peptic ulcer diseases, and bleeding, especially with long term use. Further, they do not ameliorate pain completely, requiring additional medications such as acetaminophen or opioid-based analgesics.

Shibaro is a mixture of purified oriental herbs consisting of Ledebouriellae Radix, Achyranthis Radix, Acanthopanacis Cortex, Cibotii Rhizoma, Glycine Semen, and Eucommiae Cortex. These herbs have been used for the treatment of diverse inflammatory conditions in Chines traditional medicine. All 6 herbs show an excellent safety profile and their anti-inflammatory and analgesic effects have been studied in both animals and humans. As such, given the excellent safety profile, anti-inflammatory and analgesic effects, Shinbaro might be ideal in the treatment of OA.

This study will investigate the efficacy and safety of Shinbaro in the treatment of hand OA in a placebo-controlled, randomized, double-blind, multi-center trial.

ELIGIBILITY:
Inclusion Criteria:

* Age of 40 years or older
* Osteoarthritis according to ACR 1990 criteria
* Mean joint visual analog pain score (VAS) > 30mm in the preceding 48 hours
* Patients who are will to participate

Exclusion Criteria:

* Any prior surgery of hand joints
* prior history of Shinbaro use
* Intra-articular injection of glucocorticosteroid or hyaluronic acid in the preceding 3 months
* Pregnancy or active breast feeding
* Prior hypersensitivity reaction to herbal medications
* AST or ALT elevation > 3 of upper normal limit
* GRF (MDRD) < 30 mg/min/1.73m2
* Nephrotic syndrome, other signficant kidney disease
* Patients who seem not to tolerate the study at investigator's discretion
* Patients who refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2013-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eun Bong Lee, MD PhD, Principal Investigator — Seoul National University College of Medicine; Jin Kyun Park, MD, Study Director — Seoul National University Hospital; Yun Jong Lee, MD PhD, Study Director — Seoul National Universty Bundang Hospital; Kichul Shin, MD PhD, Study Director — SMG-SNU Boramae Medical Center
Locations (3):
- South Korea (3):
  - Seoul National Univ. Bundang Hospital, Bundang, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Seoul
  - SMG-SNU Boramae Medical Center, Seoul, Seoul

REFERENCES:
- [Background] Kloppenburg M. Hand osteoarthritis-nonpharmacological and pharmacological treatments. Nat Rev Rheumatol. 2014 Apr;10(4):242-51. doi: 10.1038/nrrheum.2013.214. Epub 2014 Jan 28. PMID 24468932
- [Background] Shin K, Kim JW, Moon KW, Yang JA, Lee EY, Song YW, Lee EB. The efficacy of diacerein in hand osteoarthritis: a double-blind, randomized, placebo-controlled study. Clin Ther. 2013 Apr;35(4):431-9. doi: 10.1016/j.clinthera.2013.02.009. Epub 2013 Mar 6. PMID 23474153
- [Background] Kim JK, Park SW, Kang JW, Kim YJ, Lee SY, Shin J, Lee S, Lee SM. Effect of GCSB-5, a Herbal Formulation, on Monosodium Iodoacetate-Induced Osteoarthritis in Rats. Evid Based Complement Alternat Med. 2012;2012:730907. doi: 10.1155/2012/730907. Epub 2012 Mar 4. PMID 22474519
- [Background] Pham T, van der Heijde D, Altman RD, Anderson JJ, Bellamy N, Hochberg M, Simon L, Strand V, Woodworth T, Dougados M. OMERACT-OARSI initiative: Osteoarthritis Research Society International set of responder criteria for osteoarthritis clinical trials revisited. Osteoarthritis Cartilage. 2004 May;12(5):389-99. doi: 10.1016/j.joca.2004.02.001. PMID 15094138
- [Background] Hochberg MC, Altman RD, April KT, Benkhalti M, Guyatt G, McGowan J, Towheed T, Welch V, Wells G, Tugwell P; American College of Rheumatology. American College of Rheumatology 2012 recommendations for the use of nonpharmacologic and pharmacologic therapies in osteoarthritis of the hand, hip, and knee. Arthritis Care Res (Hoboken). 2012 Apr;64(4):465-74. doi: 10.1002/acr.21596. PMID 22563589
- [Background] Park YG, Ha CW, Han CD, Bin SI, Kim HC, Jung YB, Lim HC. A prospective, randomized, double-blind, multicenter comparative study on the safety and efficacy of Celecoxib and GCSB-5, dried extracts of six herbs, for the treatment of osteoarthritis of knee joint. J Ethnopharmacol. 2013 Oct 7;149(3):816-24. doi: 10.1016/j.jep.2013.08.008. Epub 2013 Aug 14. PMID 23954277
- [Background] Coxib and traditional NSAID Trialists' (CNT) Collaboration; Bhala N, Emberson J, Merhi A, Abramson S, Arber N, Baron JA, Bombardier C, Cannon C, Farkouh ME, FitzGerald GA, Goss P, Halls H, Hawk E, Hawkey C, Hennekens C, Hochberg M, Holland LE, Kearney PM, Laine L, Lanas A, Lance P, Laupacis A, Oates J, Patrono C, Schnitzer TJ, Solomon S, Tugwell P, Wilson K, Wittes J, Baigent C. Vascular and upper gastrointestinal effects of non-steroidal anti-inflammatory drugs: meta-analyses of individual participant data from randomised trials. Lancet. 2013 Aug 31;382(9894):769-79. doi: 10.1016/S0140-6736(13)60900-9. Epub 2013 May 30. PMID 23726390
- [Derived] Park JK, Shin K, Kang EH, Ha YJ, Lee YJ, Lee KH, Lee EY, Song YW, Choi Y, Lee EB. Efficacy and Tolerability of GCSB-5 for Hand Osteoarthritis: A Randomized, Controlled Trial. Clin Ther. 2016 Aug;38(8):1858-1868.e2. doi: 10.1016/j.clinthera.2016.06.016. Epub 2016 Jul 21. PMID 27449412

RESULTS

PARTICIPANT FLOW:
Groups:
- Shinbaro: Shinbaro, 2 capsules (300mg), twice daily, for 12 weeks
  Shinbaro
- Placebo: Placebo 2 capsules, twice daily, for 12 weeks.
  Placebo
Period: Overall Study
Arm/Group | Shinbaro | Placebo
Started | 110 | 110
Week 4 | 106 | 102
Week 8 | 98 | 99
Week 12 | 97 | 96
Week 16 | 96 | 94
Completed | 96 | 94
Not Completed | 14 | 16
Not completed — Adverse Event | 0 | 3
Not completed — Lack of Efficacy | 3 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 8 | 3
Not completed — uncertain allocation | 1 | 3
Not completed — incomplete data | 0 | 1

BASELINE CHARACTERISTICS:
Population: 1 patients in the Shinbaro group (n=110) and 3 in the placebo group (n=110) did not receive the allocated intervention as they withdrew immediately after randomization. Also, information on 1 patient in the placebo group was not complete leading to drop out.
Groups:
- Shinbaro: Shinbaro, 2 capsules (300mg), twice daily, for 12 weeks
  observation for 4 weeks
- Placebo: Placebo 2 capsules, twice daily, for 12 weeks.
  observation for 4 weeks
- Total: Total of all reporting groups
Arm/Group | Shinbaro | Placebo | Total
Number analyzed (Participants) | 109 | 106 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (7.2) | 59.4 (8.0) | 60.1 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 98 | 198
  Male | 9 | 8 | 17
Weight [Mean (Standard Deviation); unit: kg] | 58.9 (7.4) | 59.0 (8.1) | 58.9 (7.7)
Height [Mean (Standard Deviation); unit: cm] | 156.7 (6.7) | 157.0 (6.0) | 156.8 (6.3)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 23.9 (2.5) | 23.9 (2.8) | 23.9 (2.6)
Duration of OA [Mean (Standard Deviation); unit: months] | 28.6 (46.8) | 31.7 (47.2) | 30.1 (46.9)
Family history of OA [Number; unit: participants]
  Yes | 30 | 25 | 55
  No | 79 | 81 | 160
AUSCAN pain (0-100) [Mean (Standard Deviation); unit: units on a scale] — Scale ranges from 0 (no pain) to 100 (the worst possible pain).
  units on a scale | 49.7 (16.7) | 48.2 (19.9) | 48.9 (18.3)
AUSCAN stiffness score (0-100) [Mean (Standard Deviation); unit: units on a scale] — Scale ranges from 0 (no stiffness) to 100 (the worst possible stiffness).
  units on a scale | 55.2 (23.8) | 60.4 (22.8) | 57.8 (23.4)
AUSCAN function score (0-100) [Mean (Standard Deviation); unit: units on a scale] — Scale ranges from 0 (no functional limitation) to 100 (the worst possible functional limitation).
  units on a scale | 47.2 (21.8) | 46.2 (23.9) | 46.6 (22.9)
Tender joint count [Mean (Standard Deviation); unit: Joint] — Number of tender joints on examination
  Joint | 7.7 (5.2) | 6.5 (5.2) | 7.1 (5.1)
Swollen joint count [Mean (Standard Deviation); unit: Joint] — Number of swollen joints on examination (i.e. number of inflammation joints)
  Joint | 0.6 (1.8) | 0.9 (2.4) | 0.8 (2.1)
Patient global assessment (1-100) [Mean (Standard Deviation); unit: units on a scale] — Patient's general condition rated by patient. The Scale ranges from 0 (excellent condition) to 100 (the worst possible condition).
  units on a scale | 49.6 (16.5) | 50.1 (16.3) | 49.9 (16.3)
Physician global assessment (1-100) [Mean (Standard Deviation); unit: units on a scale] — Patient's general condition rated by physician The Scale ranges from 0 (excellent condition) to 100 (the worst possible condition).
  units on a scale | 43.1 (11.1) | 41.5 (13.0) | 42.3 (12.1)
Erythrocyte sedimentation rate (ESR) [Mean (Standard Deviation); unit: mm/hr] — higher ESR reflects higher degree of systemic inflammation
  mm/hr | 14.2 (14.6) | 13.3 (10.0) | 13.8 (12.5)
C-reactive protein (CRP) [Mean (Standard Deviation); unit: mg/dL] — Higher CRP reflects higher systemic inflammation
  mg/dL | 0.09 (0.11) | 0.12 (0.26) | 0.10 (0.20)
Acetaminophen [Number; unit: participants] — Number of participants who were taking acetaminophen for pain management at baseline.
  participants
    yes | 9 | 10 | 19
    no | 100 | 96 | 196
Tramadol [Number; unit: participants] — Number of participants who were taking tramadol for pain management at baseline
  participants
    Yes | 8 | 11 | 19
    no | 101 | 95 | 196
NSAIDs [Number; unit: participants] — Number of participants who were taking NSAIDs for pain management at baseline
  participants
    yes | 36 | 36 | 72
    no | 73 | 70 | 143
Glucosamine [Number; unit: participants] — Number of participants who were taking glucosamine for pain management at baseline
  participants
    yes | 14 | 13 | 27
    no | 95 | 93 | 188
Diacerin [Number; unit: participants] — Number of participants who were taking Diacerin for pain management at baseline
  participants
    yes | 5 | 3 | 8
    no | 104 | 103 | 207
Others [Number; unit: participants] — Number of participants who were taking other OA medications for pain management at baseline.
  Others .. medications for OA, not mentioned above.
  participants
    yes | 1 | 3 | 4
    no | 108 | 103 | 211

OUTCOME MEASURES:

1. Primary Outcome: AUSCAN Pain Change at 4 Weeks From Baseline
Description: Change in AUSCAN pain score at 4 weeks from baseline = Pain at 4 weeks (0-100) - Pain at baseline (0-100).
  AUSCAN Pain scale ranges from 0 (no pain) to 100 (worst possible pain).
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline and 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
units on a scale | -9.0 [-23.6 to -0.4] | -2.2 [-16.6 to 6.0]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Assuming that an improvement in AUSCAN pain score of >10 is clinically meaningful, and assuming an alpha level of 0.05 (two-tailed), a power of 0.80, and a dropout rate of 20%, the sample size calculation revealed that 220 patients should be enrolled; Test type: Superiority or Other; p = 0.014, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: AUSCAN Pain Score at 8 Weeks From Baseline
Description: Change in AUSCAN pain score at 8 weeks from baseline = Pain at 8 weeks (0-100)- Pain at baseline (0-100). AUSCAN Pain scale ranges from 0 (no pain) to 100 (worst possible pain).
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline, 8 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
units on a scale | -13.4 [-26.2 to 0.0] | -2.2 [-17.4 to 4.8]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.011, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: AUSCAN Pain Score at 12 Weeks From Baseline
Description: Change in AUSCAN pain score at 12 weeks from baseline = Pain at 12 weeks (0-100)- Pain at baseline (0-100). AUSCAN Pain scale ranges from 0 (no pain) to 100 (worst possible pain).
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline, 12 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
units on a scale | -14.6 [-30.4 to 0.0] | -8.0 [-25.0 to 7.8]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.053, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: AUSCAN Pain Score at 16 Weeks From Baseline
Description: Change in AUSCAN pain score at 16 weeks from baseline = Pain at 16 weeks (0-100)- Pain at baseline (0-100). AUSCAN Pain scale ranges from 0 (no pain) to 100 (worst possible pain).
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline and 16 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
units on a scale | -15.6 [-28.2 to 0.0] | -4.4 [-24.8 to 7.2]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.014, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: AUSCAN Stiffness at 4 Weeks Change From Baseline
Description: Change in AUSCAN stiffness score at 4 weeks from baseline = Stiffness at 4 weeks (0-100)- Stiffness at baseline (0-100). AUSCAN Stiffness scale ranges from 0 (no stiffness) to 100 (worst possible stiffness).
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline and 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
units on a scale | -9.0 [-22.0 to 3.0] | -6.0 [-23.0 to 6.0]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.728, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: AUSCAN Stiffness at 8 Weeks Change From Baseline
Description: Change in AUSCAN stiffness score at 8 weeks from baseline = Stiffness at 8 weeks (0-100)- Stiffness at baseline (0-100). AUSCAN Stiffness scale ranges from 0 (no stiffness) to 100 (worst possible stiffness).
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: baseline and 8 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
units on a scale | -12.0 [-28 to 2] | -6 [-27 to 4.0]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.229, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: AUSCAN Stiffness at 12 Weeks Change From Baseline
Description: Change in AUSCAN stiffness score at 12 weeks from baseline = Stiffness at 12 weeks (0-100)- Stiffness at baseline (0-100). AUSCAN Stiffness scale ranges from 0 (no stiffness) to 100 (worst possible stiffness).
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Basline and 12 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
units on a scale | -14.0 [-36.0 to 0] | -11.0 [-29.8 to 5]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.194, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: AUSCAN Stiffness at 16 Weeks Change From Baseline
Description: Change in AUSCAN stiffness score at 16 weeks from baseline = Stiffness at 16 weeks (0-100)- Stiffness at baseline (0-100). AUSCAN Stiffness scale ranges from 0 (no stiffness) to 100 (worst possible stiffness).
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline, 16 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
units on a scale | -10.0 [-27.0 to 2.0] | -8.0 [-27 to 5.5]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.347, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: AUSCAN Function Change at 4 Weeks From Baseline
Description: Change in AUSCAN function score at 4 weeks from baseline = Function score at 4 weeks (0-100)- Function score at baseline (0-100). AUSCAN Function score scale ranges from 0 (no functional limitation) to 100 (worst possible functional limitation).
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Basline and 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
units on a scale | -6.8 [-18.9 to 3.6] | -3.7 [-13.7 to 6.8]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.122, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: AUSCAN Function Change at 8 Weeks From Baseline
Description: Change in AUSCAN function score at 8 weeks from baseline = Function score at 8 weeks (0-100)- Function score at baseline (0-100). AUSCAN Function score scale ranges from 0 (no functional limitation) to 100 (worst possible functional limitation).
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline and 8 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
units on a scale | -9.7 [-26.9 to 2.6] | -4.8 [-18.6 to 7.7]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.097, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: AUSCAN Function Change at 12 Weeks From Baseline
Description: Change in AUSCAN function score at 12 weeks from baseline = Function score at 12 weeks (0-100)- Function score at baseline (0-100). AUSCAN Function score scale ranges from 0 (no functional limitation) to 100 (worst possible functional limitation).
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline and 12 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
units on a scale | -11 [-27.8 to 0.8] | -2.9 [-18.7 to 9.1]

12. Secondary Outcome: AUSCAN Function Change at 16 Weeks From Baseline
Description: Change in AUSCAN function score at 16 weeks from baseline = Function score at 16 weeks (0-100)- Function score at baseline (0-100). AUSCAN Function score scale ranges from 0 (no functional limitation) to 100 (worst possible functional limitation).
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline and 16 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
units on a scale | -9.9 [-28.7 to 1.8] | -4.8 [-18.7 to 9.1]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.050, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Patient Global Assessment, Change From Baseline
Description: Change in Patient global assessment (PGA) at 4 weeks from baseline = PGA at 4 weeks (0-100)- PGA score at baseline (0-100). PGA scale ranges from 0 (excellent condition) to 100 (worst possible worse possible condition).
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline and 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
units on a scale | -9.0 [-24.0 to 2.0] | -3.0 [-15.0 to 6.0]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.031, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Patient Global Assessment, Change From Baseline
Description: Change in Patient global assessment (PGA) at 8 weeks from baseline = PGA at 8 weeks (0-100)- PGA score at baseline (0-100). PGA scale ranges from 0 (excellent condition) to 100 (worst possible worse possible condition).
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline and 8 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
units on a scale | -10.0 [-24.5 to 0] | -6.0 [-18.0 to 12]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.021, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Patient Global Assessment, Change From Baseline
Description: Change in Patient global assessment (PGA) at 12 weeks from baseline = PGA at 12 weeks (0-100)- PGA score at baseline (0-100). GPA scale ranges from 0 (excellent condition) to 100 (worst possible worse possible condition).
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline and 12 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
units on a scale | -11.0 [-30.0 to 1.0] | -6.0 [-24.0 to 6.0]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.049, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Patient Global Assessment, Change From Baseline
Description: Change in Patient global assessment (PGA) at 16 weeks from baseline = PGA at 16 weeks (0-100)- PGA score at baseline (0-100). PGA scale ranges from 0 (excellent condition) to 100 (worst possible worse possible condition).
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline and 16 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
units on a scale | -10.0 [-29.0 to 3.0] | -8.5 [-21.0 to 9.0]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.221, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Physician Global Assessment, Change From Baseline
Description: Change in Physician global assessment (PhGA) at 4 weeks from baseline = PhGA at 4 weeks (0-100)- PhGA score at baseline (0-100). GPA scale ranges from 0 (excellent condition) to 100 (worst possible worse possible condition).
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: baseline and 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
units on a scale | -12 [-21.0 to 0] | -7.0 [-19.0 to 1.0]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.174, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Physician Global Assessment, Change From Baseline
Description: Change in Physician global assessment (PhGA) at 8 weeks from baseline = PhGA at 8 weeks (0-100)- PhGA score at baseline (0-100). PhGA scale ranges from 0 (excellent condition) to 100 (worst possible worse possible condition).
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline and 8 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
units on a scale | -16.0 [-26.0 to -4.0] | -11.5 [-25.3 to 0.0]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.124, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Physician Global Assessment, Change From Baseline
Description: Change in Physician global assessment (PhGA) at 12 weeks from baseline = PhGA at 12 weeks (0-100)- PhGA score at baseline (0-100). PhGA scale ranges from 0 (excellent condition) to 100 (worst possible worse possible condition).
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline and 12 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
units on a scale | -19.0 [-29.0 to -5.0] | -13 [-27.0 to 0.0]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.128, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Physician Global Assessment, Change From Baseline
Description: Change in Physician global assessment (PhGA) at 16 weeks from baseline = PhGA at 16 weeks (0-100)- PhGA score at baseline (0-100). PhGA scale ranges from 0 (excellent condition) to 100 (worst possible worse possible condition).
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline and 16 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
units on a scale | -12 [-23.5 to 0] | -6.5 [-20.0 to 1.0]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.126, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Tender Joint Count, Change From Baseline
Description: Change in Tender joint count (TJC) at 4 weeks from baseline = TJC at 4 weeks - TJC at baseline..
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline and 4 weeks
Measure: Median (Inter-Quartile Range); unit: joints
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
joints | -1 [-4 to 0] | 0 [-3.0 to 1.0]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.042, Wilcoxon (Mann-Whitney)

22. Secondary Outcome: Tender Joint Count, Change From Baseline
Description: Change in Tender joint count (TJC) at 8 weeks from baseline = TJC at 8 weeks - TJC at baseline..
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline and 8 weeks
Measure: Median (Inter-Quartile Range); unit: Joints
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
Joints | -1.0 [-4.0 to 0] | -1.0 [-5 to 0]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.660, Wilcoxon (Mann-Whitney)

23. Secondary Outcome: Tender Joint Count, Change From Baseline
Description: Change in Tender joint count (TJC) at 12 weeks from baseline = TJC at 12 weeks - TJC at baseline..
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline and 12 weeks
Measure: Median (Inter-Quartile Range); unit: joints
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
joints | -2.0 [-5.0 to 0] | -1.0 [-4.0 to 0]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.006, Wilcoxon (Mann-Whitney)

24. Secondary Outcome: Tender Joint Count, Change From Baseline
Description: Change in Tender joint count (TJC) at 16 weeks from baseline = TJC at 16 weeks - TJC at baseline..
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline and 16 weeks
Measure: Median (Inter-Quartile Range); unit: joints
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
joints | -2.0 [-5.0 to 1.0] | -1.0 [-5.0 to 1.0]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.186, Wilcoxon (Mann-Whitney)

25. Secondary Outcome: Swollen Joint Count, Change From Baseline
Description: Change in Swollen joint count (SJC) at 4 weeks from baseline = SJC at 4 weeks - TJC at baseline..
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline and 4 weeks
Measure: Median (Inter-Quartile Range); unit: Joints
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
Joints | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.493, Wilcoxon (Mann-Whitney)

26. Secondary Outcome: Swollen Joint Count, Change From Baseline
Description: Change in Swollen joint count (SJC) at 8 weeks from baseline = SJC at 8 weeks - TJC at baseline..
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline and 8 weeks
Measure: Median (Inter-Quartile Range); unit: Joints
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
Joints | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.062, Wilcoxon (Mann-Whitney)

27. Secondary Outcome: Swollen Joint Count, Change From Baseline
Description: Change in Swollen joint count (SJC) at 12 weeks from baseline = SJC at 12 weeks - TJC at baseline..
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline and 12 weeks
Measure: Median (Inter-Quartile Range); unit: Joints
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
Joints | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.604, Wilcoxon (Mann-Whitney)

28. Secondary Outcome: Swollen Joint Count, Change From Baseline
Description: Change in Swollen joint count (SJC) at 16 weeks from baseline = SJC at 16 weeks - TJC at baseline..
  * Negative value means improvement from baseline
  * Positive value means deterioration from baseline
Time Frame: Baseline and 16 weeks
Measure: Median (Inter-Quartile Range); unit: Joints
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
Joints | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.252, Wilcoxon (Mann-Whitney)

29. Secondary Outcome: Acetaminophen Rescue
Description: yes = AAP rescue use, no = no AAP rescue use
Time Frame: Baseline 4 weeks
Measure: Number; unit: participants
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
participants
  yes | 7 | 4
  no | 102 | 102
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.378, Chi-squared

30. Secondary Outcome: Acetaminophen Rescue
Description: yes = AAP rescue use, no = no AAP rescue use
Time Frame: 4 weeks and 8 weeks
Measure: Number; unit: participants
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
participants
  yes | 10 | 7
  no | 99 | 99
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.485, Chi-squared

31. Secondary Outcome: Acetaminophen Rescue
Description: yes = AAP rescue use, no = no AAP rescue use
Time Frame: 8 weeks and 12 weeks
Measure: Number; unit: participants
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
participants
  yes | 4 | 4
  no | 105 | 102
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 1.000, Fisher Exact

32. Secondary Outcome: Acetaminophen Rescue
Description: yes = AAP rescue use, no = no AAP rescue use
Time Frame: 12 weeks and 16 weeks
Measure: Number; unit: participants
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
participants
  yes | 4 | 2
  no | 105 | 104
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.683, Fisher Exact

33. Secondary Outcome: Number of OMERACT-OARSI Responder
Description: Outcome Measures in Rheumatology-Osteoarthritis Research Society International (OMERACT-OARSI) Number of patients who met OMERACT-OARSI criteria = significant clinical improvement in osteoarthritis symptom after treatment
Time Frame: Baseline and 4 weeks
Measure: Number; unit: participants
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
participants
  Responder | 48 | 32
  Nonresponder | 61 | 74
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.036, Chi-squared

34. Secondary Outcome: Number of OMERACT-OARSI Responder
Description: Number of patients who met OMERACT-OARSI criteria = significant clinical improvement in osteoarthritis symptom after treatment
Time Frame: Baseline and 8 weeks
Measure: Number; unit: participants
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
participants
  responder | 56 | 38
  nonresponder | 53 | 68
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.022, Chi-squared

35. Secondary Outcome: Number of OMERACT-OARSI Responder
Description: as for outcome 34
Time Frame: Baseline and 12 weeks
Measure: Number; unit: participants
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
participants
  responder | 62 | 43
  nonresponder | 47 | 63
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.017, Chi-squared

36. Secondary Outcome: Number of OMERACT-OARSI Responder
Description: as for outcome 34
Time Frame: Baselie and 16 weeks
Measure: Number; unit: participants
Arm/Group | Shinbaro | Placebo
Number analyzed (Participants) | 109 | 106
participants | 55 | 40
Statistical Analysis 1: Comparison: Shinbaro vs Placebo; Test type: Superiority or Other; p = 0.060, Chi-squared

ADVERSE EVENTS:
Time Frame: Any event between randomization (week 0) and study end (week 16)
Groups:
- Shinbaro: GCSB-5 (Shinbaro), 2 capsules (300mg), twice daily, for 12 weeks
  observation for 4 weeks
Arm/Group | Shinbaro | Placebo
Serious Adverse Events (participants affected / at risk) | 1/109 | 4/106
Other Adverse Events (participants affected / at risk) | 55/109 | 45/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Shinbaro (N=109) | Placebo (N=106)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 — Fracture
Surgery (General disorders) | 1 | 1 — Surgery
Skin rash (Musculoskeletal and connective tissue disorders) | 0 | 1
liver function abnormality (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Shinbaro (N=109) | Placebo (N=106)
Headache (Nervous system disorders) | 4 | 3
Dizziness (Nervous system disorders) | 1 | 2
Paresthesia (Nervous system disorders) | 2 | 4
Skin rash (Skin and subcutaneous tissue disorders) | 10 | 12
Nausea (Gastrointestinal disorders) | 9 | 10
Abdominal discomfort (Gastrointestinal disorders) | 18 | 13
Diarrhea (Gastrointestinal disorders) | 1 | 2
Liver function change (Hepatobiliary disorders) | 8 | 8
Leukopenia (Blood and lymphatic system disorders) | 11 | 8
Anemia (Blood and lymphatic system disorders) | 2 | 4
Upper respiratory infection (Immune system disorders) | 16 | 5
Zoster (Immune system disorders) | 0 | 1
Visual floater (Eye disorders) | 1 | 0
Depressive mood (Psychiatric disorders) | 0 | 1
insomnia (Psychiatric disorders) | 0 | 3
Surgery (Surgical and medical procedures) | 1 | 1
Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No